CLINICAL TRIAL: NCT05629559
Title: An Open-Label, Phase 1/2a Trial of Gene Therapy 4D-310 in Adults With Fabry Disease and Cardiac Involvement
Brief Title: 4D-310 in Adults With Fabry Disease and Cardiac Involvement
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4D-310-C002
Record Dates: First submitted 2022-11-04; First posted 2022-11-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Fabry Disease
Keywords: Lysosomal Storage Diseases; Nervous System Brain Diseases; Metabolic; Inborn Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cerebral Small Vessel Diseases; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Genetic Diseases; X-Linked; Inborn; Metabolic Diseases; Lipid Metabolism Disorders; Sphingolipidoses; Metabolism; Inborn Errors; Lipidoses; Lipid Metabolism
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases; Central Nervous System Diseases; Nervous System Diseases; Cerebral Small Vessel Diseases; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Genetic Diseases, Inborn; Metabolic Diseases; Lipid Metabolism Disorders; Sphingolipidoses; Lipidoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 4D-310 Dose Level -1 (Experimental): Single IV administration of 4D-310 Dose Level -1
  Interventions: Biological: 4D-310
- 4D-310 Dose Level 2 (Experimental): Single IV administration of 4D-310 Dose Level 2
  Interventions: Biological: 4D-310
- 4D-310 Dose Level 3 (Experimental): Single IV administration of 4D-310 at Dose Level 3
  Interventions: Biological: 4D-310
- 4D-310 Dose Level 1 (No longer enrolling) (Experimental): No longer enrolling - Single IV administration of 4D-310 at Dose Level 1
  Interventions: Biological: 4D-310

INTERVENTIONS:
Biological: 4D-310 — Single IV administration of 4D-310

SUMMARY:
This is a prospective multicenter, open-label, dose-escalation trial to assess the safety, tolerability, and pharmacodynamics of 4D-310 following a single IV administration. The study population is comprised of adult males and females with Fabry Disease and cardiac involvement

DETAILED DESCRIPTION:
This is a prospective multicenter, open-label, dose-escalation trial to assess the safety, tolerability, and pharmacodynamics of 4D-310 following a single IV administration. The study population is comprised of adult males and females with Fabry Disease and cardiac involvement

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 to ≤65 years of age
2. Pathogenic GLA mutation consistent with Fabry Disease
3. Confirmed diagnosis of classic or late-onset Fabry disease with cardiac involvement
4. Intolerant of ERT, unable or unwilling to receive ERT, or progressive disease despite ERT or migalastat
5. Individuals receiving ERT, must be on a stable dose for at least 6 months
6. Agree to use highly effective contraception

Exclusion Criteria:

1. Presence of pre-existing antibodies to 4D-310 capsid or to AGA
2. eGFR <65 mL/min/1.73 m2
3. Undergone kidney transplantation or currently on hemodialysis or peritoneal dialysis
4. HIV, active or chronic hepatitis B or C,
5. Evidence of liver disease, severe pulmonary disease or diabetes with poor glycemic control
6. History of stroke or transient ischemic attack within the last 12 months, or other significant thromboembolic disease history (e.g. pulmonary embolism)
7. Contraindication to systemic corticosteroid therapy or immunosuppressive therapy
8. Chronic steroid use, defined as ≥ 3 months of oral corticosteroid use within the last 12 months.
9. Moderately severe to severe cardiovascular disease or uncontrolled hypertension
10. Left ventricular ejection fraction of <45% on echocardiogram (ECHO)
11. Currently receiving investigational drug, device or therapy or having ever received gene therapy
12. History of infusion related response to ERT or any adverse reaction leading to ERT discontinuation
13. History of cancer within 2 years (exceptions include non-melanoma skin cancer, localized prostate cancer treated with curative intent)
14. Pregnant or breast-feeding

Note: Other inclusion and exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 1 year
  Incidence and severity of adverse events following a single IV dose of 4D-310intravenous (IV) dose

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Cohen, MD, Study Director — 4D Molecular Therapeutics
Locations (4):
- Australia (3):
  - Royal Melbourne Hospital, Melbourne
  - Royal Perth Hospital, Perth
  - Westmead Hospital, Westmead
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No